CLINICAL TRIAL: NCT00461123
Title: A Randomized, Double-blind, Parallel Group Prospective Pilot Study to Assess the Effect of Vardenafil on Clinical Outcome and on Procedure Duration After Green Light Laser-ablation of the Prostate Gland for Therapy of Benign Prostate Hypertrophy (BPH)
Brief Title: Vardenafil in Greenlight(TM) Laser Surgery of Benign Prostate Hypertrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12496; 2006-004633-15 (EudraCT Number)
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Results first posted 2010-01-21 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Prostatic Hypertrophy, Benign
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil (Levitra, BAY38-9456) (Experimental): One tablet vardenafil 10 mg with a glass of water the evening before ablation of prostate; the second dose (vardenafil 20 mg) with a glass of water approximately one hour before Greenlight(TM) laser ablation of prostate commenced.
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)
- Placebo (Placebo Comparator): One placebo tablet with a glass of water the evening before ablation of prostate; the second placebo dose with a glass of water approximately one hour before Greenlight(TM) laser ablation of prostate commenced.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — One tablet vardenafil 10 mg with a glass of water the evening before ablation of prostate; the second dose (vardenafil 20 mg) with a glass of water approximately one hour before Greenlight(TM) laser ablation of prostate commenced.
  Arms: Vardenafil (Levitra, BAY38-9456)
Drug: Placebo — One placebo tablet with a glass of water the evening before ablation of prostate; the second placebo dose with a glass of water approximately one hour before Greenlight(TM) laser ablation of prostate commenced.
  Arms: Placebo

SUMMARY:
The greenlight laser has an absorption maximum which is exactly the same as for hemoglobin. In the presence of hemoglobin, its application causes vaporization of the tissue and this effect depends on the concentration of hemoglobin in the respective tissue. Therefore, increase of blood-flow in the tissue (here: prostate gland) should exert better efficacy of the laser application and consequently shortening of the required duration of laser application.

ELIGIBILITY:
Inclusion Criteria:

* Men with benign prostate hypertrophy requiring surgical treatment
* Age up to 80 years
* Documented, dated, written Informed Consent
* Anesthesiologists agreement with swallowing 1 tablet one hour prior surgery

Exclusion Criteria:

* Any unstable medical, psychiatric, or substance abuse disorder
* History of previous prostatectomy
* Patients suspect of prostate cancer
* Hereditary degenerative retinal disorder
* History of previous Non-arteric Anterior Ischemic Optic Neuropathy (NAION) episode or unilateral vision impairment
* Any cardiovascular condition
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Uncontrolled atrial fibrillation/flutter at screening
* Severe chronic or acute liver disease
* Chronic hematological disease which may lead to priapism
* Bleeding disorder
* Significant active peptic ulceration
* Resting hypotension
* History of positive test for Hepatitis B surface antigen or Hepatitis C
* Symptomatic postural hypotension within 6 months of Visit 1
* Patients who subjectively or in the opinion of the investigator did not tolerate the initial dose of study medication well
* Subjects who are taking nitrates or nitric oxide donors
* Subjects who are taking androgens or anti-androgens
* Subjects who are taking potent inhibitors of cytochrome P4503A4
* Subjects who have received any investigational drug within 30 days of Visit 1
* Using of alpha-blockers during two days prior to first dosing of study medication and after ablation of prostate
* Use of inhibitors of 5-alpha reductase after ablation of prostate
* Subjects with serum creatinine clearance <30.0 mL/min
* Elevation of Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) >3 times the upper limit of normal
* Subjects with known hypersensitivity to Vardenafil
* Subjects who are illiterate or unable to understand subject diaries
* Subjects who would be non-compliant with the study visit schedule

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Click here and search for Bayer Product information by EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started on 19 March 2007 and the last study visit occurred on 02 June 2008. The study was conducted at one center, a university clinic in Germany.
Pre-assignment Details: Number of subjects enrolled, randomized and exposed to at least one dose (safety population): 50. Number of subjects who had undergone surgery, whose type of surgery (Greenlight(TM) laser-ablation) had not changed, energy consumption during surgery reported and who had taken the second dose on the day of surgery (intent-to-treat population): 44
Groups:
- Vardenafil (Levitra, BAY38-9456): One tablet vardenafil 10 mg with a glass of water the evening before ablation of prostate; the second dose (vardenafil 20 mg) with a glass of water approximately one hour before GreenlightTM laser ablation of prostate commences.
- Placebo: One placebo tablet with a glass of water the evening before ablation of prostate; the second placebo dose with a glass of water approximately one hour before GreenlightTM laser ablation of prostate commences
Period: Overall Study
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Started | 25 | 25
Completed | 19 | 19
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.5) | 65.9 (7.9) | 65.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted Least Squared (LS) Means of Peak Urinary Flow (Qmax) at 3 Months After Surgery or Last Observation Carried Forward (LOCF)
Description: Baseline (pre-surgery Day -1) adjusted least squares (LS)-means at 3 months after surgery (Day +90, last observation carried forward (LOCF)) in peak urinary flow.
Time Frame: baseline and up to 3 months after surgery
Population: The intent-to-treat (ITT) population includes participants with baseline and post-baseline measurement of peak urinary flow; imputation technique: last post-baseline observation carried forward (LOCF). The ITT population is not identical to the number of subjects who "completed" the study, as displayed under Participants Flow.
Measure: Mean (Standard Deviation); unit: milliliter per second (mL/s)
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 19 | 18
milliliter per second (mL/s)
  baseline mean | 8.3 (4.08) | 9.4 (5.69)
  Day +90 or LOCF mean | 23.1 (10.60) | 25.7 (7.90)
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; null hypothesis: mean of Vardenafil group equals mean of Placebo group at day +90; Test type: Superiority or Other; p = 0.5248, ANCOVA; Analysis of covariance (ANCOVA), baseline as covariate, treatment as fixed factor; Mean Difference (Final Values) = 1.93, 95% CI [-4.18 to 8.05] — Difference of least squares (LS) means (Placebo minus Vardenafil)

2. Secondary Outcome: Baseline-adjusted Least Squared (LS) Means of International Prostate Symptom Score (IPSS) Total Score at 3 Months After Surgery or Last Observation Carried Forward (LOCF)
Description: Baseline (pre-surgery Day -1) adjusted LS-means at 3 months after surgery (Day +90, LOCF) in IPSS total score. IPSS is a questionnaire on benign prostate hyperplasia, including seven 6-point items on symptoms and one 7-point item on quality of life. Total score: sum of items 1 through 7; minimum: 0 (best); maximum: 41 (worst).
Time Frame: baseline and up to 3 months after surgery
Population: The intent-to-treat (ITT) population includes participants with baseline and post-baseline measurement of International Prostate Symptom Score (IPSS) total score; imputation technique: last post-baseline observation carried forward (LOCF). The ITT population is not identical to the number of subjects who "completed" the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 20 | 19
scores on a scale
  baseline mean | 19.1 (5.92) | 19.7 (5.83)
  Day +90 or LOCF mean | 6.9 (4.25) | 6.7 (6.03)
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; null hypothesis: mean of Vardenafil group equals mean of Placebo group at day +90; Test type: Superiority or Other; p = 0.8700, ANCOVA; Analysis of covariance (ANCOVA), baseline as covariate, treatment as fixed factor; Mean Difference (Final Values) = -0.27, 95% CI [-3.58 to 3.04] — Difference of LS means (Placebo minus Vardenafil)

3. Secondary Outcome: Baseline-adjusted Least Squared (LS) Means of Post-void Residual (PVR) Volume at 3 Months After Surgery or Last Observation Carried Forward (LOCF)
Description: Baseline (pre-surgery Day -1) adjusted LS-means at 3 months after surgery (Day +90, last observation carried forward (LOCF)) in PVR volume. PVR is the amount of urine left in the bladder after a person has passed urine.
Time Frame: baseline and up to 3 months after surgery
Population: The intent-to-treat (ITT) population includes participants with baseline and post-baseline measurement of post-void residual (PVR) volume; imputation technique: last post-baseline observation carried forward (LOCF). The ITT population is not identical to the number of subjects who "completed" the study.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 18 | 17
milliliter (mL)
  baseline mean | 139.3 (116.43) | 117.4 (81.42)
  Day +90 or LOCF mean | 18.7 (23.55) | 22.5 (18.34)
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; null hypothesis: mean of Vardenafil group equals mean of Placebo group at day +90; Test type: Superiority or Other; p = 0.4162, ANCOVA; Analysis of covariance (ANCOVA), baseline as covariate, treatment as fixed factor; Mean Difference (Final Values) = 5.57, 95% CI [-8.21 to 19.35] — Difference of LS means (Placebo minus Vardenafil)

4. Secondary Outcome: Baseline-adjusted Least Squared (LS) Means of the Number of Urinary Incontinence Episodes Per Week at 3 Months After Surgery or Last Observation Carried Forward (LOCF)
Description: Baseline (pre-surgery Day -1) adjusted LS-means at 3 months after surgery (Day +90, last observation carried forward (LOCF)) in the number of incontinence episodes. Urinary incontinence is an involuntary excretion (passing) of urine. Urinary incontinence episodes were collected in the patient diary.
Time Frame: baseline and up to 3 months after surgery
Population: The intent-to-treat (ITT) population includes participants with baseline and post-baseline documentation of number of incontinence episodes per week; imputation technique: last post-baseline observation carried forward (LOCF). The ITT population is not identical to the number of subjects who "completed" the study.
Measure: Mean (Standard Deviation); unit: urinary incontinence episodes
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 17 | 18
urinary incontinence episodes
  baseline mean | 8.4 (25.71) | 0.0 (0.00)
  Day +90 or LOCF mean | 7.1 (13.42) | 0.4 (1.42)
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; null hypothesis: mean of Vardenafil group equals mean of Placebo group at day +90; Test type: Superiority or Other; p = 0.0588, ANCOVA; Analysis of covariance (ANCOVA), baseline as covariate, treatment as fixed factor; Mean Difference (Final Values) = -6.50, 95% CI [-13.25 to 0.26] — Difference of LS means (Placebo minus Vardenafil)

5. Secondary Outcome: Duration of Surgery
Description: Duration of prostate laser ablation, i.e. Greenlight(TM) laser surgery.
Time Frame: on the day of surgery, without any further allowable time window
Population: The intent-to-treat (ITT) population includes participants with baseline and post-baseline measurement of duration of surgery; imputation technique: last post-baseline observation carried forward (LOCF). The ITT population is not identical to the number of subjects who "completed" the study.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 23 | 21
minutes | 75.1 (36.5) | 72.5 (25.8)
Statistical Analysis 1: Comparison: Vardenafil (Levitra, BAY38-9456) vs Placebo; null hypothesis: mean of Vardenafil group equals mean of Placebo group; Test type: Superiority or Other; p = 0.7878, ANCOVA; Analysis of variance (ANOVA), treatment as fixed factor; Mean Difference (Net) = -2.61, 95% CI [-22.03 to 16.82] — Difference of LS means (Placebo minus Vardenafil)

ADVERSE EVENTS:
Arm/Group | Vardenafil (Levitra, BAY38-9456) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 2/25
Other Adverse Events (participants affected / at risk) | 2/25 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil (Levitra, BAY38-9456) (N=25) | Placebo (N=25)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil (Levitra, BAY38-9456) (N=25) | Placebo (N=25)
Pyrexia (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No